CLINICAL TRIAL: NCT06294483
Title: Comparison of Clinical Features, Hematological Indices and Disease Activity Between Early-onset and Late-onset Patients With Systemic Lupus Erythematosus.
Brief Title: Comparison Between Early-onset and Late-onset Patients With Systemic Lupus Erythematosus.
Status: Enrolling by invitation | Type: Observational
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, Esraa Ali kobsy, : internal medicine resident in Sohag university hospital, Sohag University
Other Study IDs: Soh-Med-24-01-09MS
Record Dates: First submitted 2024-02-04; First posted 2024-03-05 (Actual); Last update posted 2024-03-05 (Actual); Status verified 2024-03

CONDITIONS: Systemic Lupus Erythematosus
MeSH Terms: conditions — Lupus Erythematosus, Systemic

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- early onset SLE: group of patients diagnosed as SLE before age of fifty years old
  Interventions: Diagnostic Test: CBC; Diagnostic Test: Antinuclear Antibody tests (ANA); Diagnostic Test: Rest of ANA profile; Diagnostic Test: C3 and C4 complement level.; Diagnostic Test: Anti phospholipid marker; Diagnostic Test: Serum creatinine and Alb/create ratio; Other: 2019 European League Against Rheumatism/American College of Rheumatology classification criteria for systemic lupus erythematosus.; Other: SLEDAI scores
- late onset SLE: Patients were diagnosed as SLE at age of fifty years old or more
  Interventions: Diagnostic Test: CBC; Diagnostic Test: Antinuclear Antibody tests (ANA); Diagnostic Test: Rest of ANA profile; Diagnostic Test: C3 and C4 complement level.; Diagnostic Test: Anti phospholipid marker; Diagnostic Test: Serum creatinine and Alb/create ratio; Other: 2019 European League Against Rheumatism/American College of Rheumatology classification criteria for systemic lupus erythematosus.; Other: SLEDAI scores

INTERVENTIONS:
Diagnostic Test: CBC — Is used to detect haematological indices (mean platelet volume, platelet lymphocyte ratio and neutrophil lymphocyte ratio) and its relation to disease activity
Diagnostic Test: Antinuclear Antibody tests (ANA) — To be tool in diagnosis of SLE
Diagnostic Test: Rest of ANA profile — As tool of diagnosis of SLE
Diagnostic Test: C3 and C4 complement level. — As method of detection of acute acivity of SLE
Diagnostic Test: Anti phospholipid marker — To detect antiphospholipid syndrome if there is sign of thrombosis
Diagnostic Test: Serum creatinine and Alb/create ratio — To detct complication of disease on kidney
Other: 2019 European League Against Rheumatism/American College of Rheumatology classification criteria for systemic lupus erythematosus. — Is criteria of diagnosis of SLE
Other: SLEDAI scores — Is score to detect the activity of disease

SUMMARY:
The present study aims to:

Compare clinical features, hematological indices and disease activity between the early-onset and late-onset patients with systemic lupus erythematosus.

Evaluate the relationship between hematological indices (mean platelet volume, platelet lymphocyte ratio and neutrophil lymphocyte ratio) and Systemic lupus erythematosus (SLE) disease manifestations and activity.

DETAILED DESCRIPTION:
This is a cross sectional study, patients with SLE will be gathered from the Internal medicine department and Rheumatology and Immunology outpatient clinic in Sohag university hospital. All patients fulfilled 2019 European League Against Rheumatism/American College of Rheumatology classification criteria for systemic lupus erythematosus.

In this study, 100 SLE patients will be classified into two groups:

Group A: early onset SLE (age at diagnosis < 50 years). Group B: late onset SLE. (age at diagnosis ≥ 50

Data collection procedure:

The following clinical data will be collected:

Clinical assessment:

Name, age, gender, smoker or ex-smoker or non-smoker, blood pressure and body mass index.

Clinical manifestations as:

Malar rash. Discoid rash. Photosensitivity. Mucocutaneous or oral ulcer. Alopecia. Raynaud's phenomena. History of deep venous thrombosis. Cutaneous vasculitis. Fever. Lupus nephritis. Arthritis. Myositis. Secondary antiphospholipid syndrome. Serositis. Pleural effusion. Renal manifestations (puffiness and lower limb edema). Neurological (headache, seizers, psychosis and Disturbed conscious level)

Hematological manifestations:

Thrombocytopenia (bleeding tendency) Anemia and Hemolytic anemia (anemic manifestation). Hypertension. Diabetes mellitus. Previous coronary event or Peripheral vascular disease.

Laboratory assessment:

1. CBC with differential WBCs count.
2. Antinuclear Antibody tests (ANA).
3. Anti-double-stranded DNA (ds DNA).
4. Anti-Sm.
5. C3 and C4 complement level.
6. Serum creatinine level.
7. Anti phospholipid marker (if needed). Each clinical data and laboratory results will be put into the SLEDAI score. The score is considered accurate and reliable. Categories of disease activity based on SLEDAI scores are as follows: no activity (SLEDAI= 0), mild activity (SLEDAI= 1-5), moderate activity (SLEDAI= 6-10), high activity (SLEDAI= 11-19) and very high activity (SLEDAI= 20).

The present study aims to:

Compare clinical features, and disease activity as SLEDAI score between the early-onset and late-onset patients with systemic lupus erythematosus.

Evaluate the relationship between hematological indices (mean platelet volume, platelet lymphocyte ratio and neutrophil lymphocyte ratio) and Systemic lupus erythematosus (SLE) disease manifestations and activity

Duration of study:

Six months after approval of the protocol by Medical Research Ethics Committee of Sohag faculty of medicine.

Inclusion criteria:

All patients fulfilled 2019 European League Against Rheumatism/American College of Rheumatology classification criteria for systemic lupus erythematosus.

Exclusion Criteria:

Patients received glucocorticoid or immunosuppressant medication. Patients presented with other chronic inflammatory diseases, infection, or other autoimmune diseases at the time of diagnosis Malignancy Pregnancy.

ELIGIBILITY:
Inclusion Criteria:

* All patients fulfilled 2019 European League Against Rheumatism/American College of Rheumatology classification criteria for systemic lupus erythematosus.

Exclusion Criteria:

* Patients received glucocorticoid or immunosuppressant medication. Patients presented with other chronic inflammatory diseases, infection, or other autoimmune diseases at the time of diagnosis Malignancy Pregnancy.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All patients fulfilled 2019 European League Against Rheumatism/American College of Rheumatology classification criteria for systemic lupus erythematosus.
  While include In this study as 100 SLE patients will be classified into two groups:
  Group A: early onset SLE (age at diagnosis < 50 years). Group B: late onset SLE. (age at diagnosis ≥ 50 years).
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2024-01-10 (Actual); Primary Completion 2024-07-30 (Estimated); Study Completion 2024-08-30 (Estimated)

PRIMARY OUTCOMES:
Evaluate the hematological indices as (mean platelet volume) of our SLE patient. | for 2 weeks after admission of patient in sohag university hospital]
  Neutrophils, lymphocytes, and platelets play important roles in the course of various diseases . In recent years, there has been a growing interest in the role of hematological indices (mean platelet volume, platelet lymphocyte ratio and neutrophil lymphocyte ratio) to estimate disease activity in some auto-immune diseases as and SLE . Neutrophil-to-lymphocyte ratio (NLR), platelet-to-lymphocyte ratio (PLR), as CBC parameters, have recently shown to be useful markers of inflammation in autoimmune and inflammatory disorders so we will do CBC for our pt to detect mean platelet volume
Evaluate the hematological indices as (neutrophil lymphocyte ratio) of our SLE patient. | for 2 weeks after admission of patient in sohag university hospital]
  Neutrophils, lymphocytes, and platelets play important roles in the course of various diseases . In recent years, there has been a growing interest in the role of hematological indices (mean platelet volume, platelet lymphocyte ratio and neutrophil lymphocyte ratio) to estimate disease activity in some auto-immune diseases as and SLE . Neutrophil-to-lymphocyte ratio (NLR), platelet-to-lymphocyte ratio (PLR), as CBC parameters, have recently shown to be useful markers of inflammation in autoimmune and inflammatory disorders so we will do CBC for our pt to detect this neutrophil lymphocyte ratio
Evaluate the hematological indices ( platelet lymphocyte ratio ) of our SLE patient. | for 2 weeks after admission of patient in sohag university hospital]
  Neutrophils, lymphocytes, and platelets play important roles in the course of various diseases . In recent years, there has been a growing interest in the role of hematological indices (mean platelet volume, platelet lymphocyte ratio and neutrophil lymphocyte ratio) to estimate disease activity in some auto-immune diseases as and SLE . Neutrophil-to-lymphocyte ratio (NLR), platelet-to-lymphocyte ratio (PLR), as CBC parameters, have recently shown to be useful markers of inflammation in autoimmune and inflammatory disorders so we will do CBC for our pt to detect platelet lymphocyte ratio
Compare the degree of disease activity between the early-onset and late-onset patients with systemic lupus erythematosus. | for 2 weeks after admission of patient in sohag university hospital]
  Each clinical data and laboratory results will be put into the SLEDAI score. The score is considered accurate and reliable. Categories of disease activity based on SLEDAI scores are as follows: no activity (SLEDAI= 0), mild activity (SLEDAI= 1-5), moderate activity (SLEDAI= 6-10), high activity (SLEDAI= 11-19) and very high activity (SLEDAI= 20).
Evaluate the correlation between hematological indices (mean platelet volume, platelet lymphocyte ratio and neutrophil lymphocyte ratio) and Systemic lupus erythematosus (SLE) disease manifestations and activity. | for 2 weeks after admission of patient in sohag university hospital
  After detection of previous outcome [ disease activity , clinical feature,haematological indices ] we will compare them to detect the correlation between them for every patient

CONTACTS AND LOCATIONS:
Locations (1):
- Sohag university hospital, Sohag, Egypt

IPD SHARING:
Plan to Share IPD: Undecided